CLINICAL TRIAL: NCT06065345
Title: BIOTRONIK- Pharmacokinetic Study of a Sirolimus Derivative-Coated Balloon (BRight DCB) in the Superficial Femoral and Proximal Popliteal Artery
Brief Title: BRight Pharmacokinetic Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik CRC Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C2304
Record Dates: First submitted 2023-09-18; First posted 2023-10-03 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BRight DCB (Experimental): Single arm study. All subjects will be treated with the BRight DCB
  Interventions: Device: BRight DCB

INTERVENTIONS:
Device: BRight DCB — The BRight Drug-Coated Percutaneous Transluminal Angioplasty (PTA) Balloon catheter (BRight DCB) is intended for dilatation of de novo lesions in native superficial femoral or popliteal arteries with a simultaneous release of drug to the vessel wall as a secondary action to reduce occurrence of a restenosis of the treated vessel segment.

SUMMARY:
The BRight PK Study is a prospective, single-arm, open-label, non-blinded, non-randomized study, which goal is to assess the pharmacokinetic profile of the BRight drug-coated balloon at different time points after the balloon deployment.

The study will enroll a maximum of 10 patients at a single site in Australia

ELIGIBILITY:
Inclusion Criteria:

1. The subject has provided written informed consent
2. The subject is willing to participate in the clinical investigation and to comply with the study procedures and follow-up visits
3. Lifestyle-limiting claudication or rest pain requiring treatment of superficial femoral (SFA) and/or proximal popliteal artery (PPA)
4. Age ≥ 18 years old
5. Rutherford-Becker Clinical Category of 2, 3 or 4
6. Target vessel reference diameter ≥5 mm and ≤ 6 mm (by visual estimation)
7. De novo lesion with >50% stenosis by operator visual estimate within the SFA and/or proximal popliteal arteries in a single limb.
8. Lesion must be located ≥ 1 cm below the Common Femoral Artery (CFA) bifurcation and terminate distally at ≥ 3 cm proximal to the knee joint (radiographic joint space).
9. Single lesion length ≤170 mm for de novo stenotic lesions, or ≤ 100 mm for occluded lesions (one long lesion or multiple serial lesions) by operator visual estimate. Notes: (1) Only 1 lesion per patient can be treated. Multiple serial lesions are allowed if they can be treated as a single lesion with a maximum of 2 balloons. (2) a non-occlusive lesion that includes a totally occluded segment along its length are eligible provided that the overall treated lesion length is ≤170 mm (with / or without an occluded segment not greater than 100 mm in length).
10. Successful guidewire crossing of lesion.
11. After pre-dilatation, the target lesion is ≤ 30% residual stenosis with no flow limiting dissection and treatable with a maximum of 2 balloons.
12. Inflow artery is patent, free from significant lesion stenosis (>50% stenosis considered significant) as confirmed by angiography.

    Note: Where required, inflow iliac arteries (common and external iliac arteries only) must be successfully treated during the index procedure. Completion angiography must confirm successful treatment of inflow disease (≤50% residual stenosis, no distal embolization, and no Grade C or greater dissection) prior to pre-dilatation of the target lesion. Drug-eluting devices are not allowed for treatment of the occluded inflow iliac arteries.
13. Patency of the popliteal segments P2 and P3 with at least 1 patent infrapopliteal run-off vessel (that may have a stenosis of less than 50% not interfering with the outflow to the pedal arch) to the ankle in continuity with the native femoropopliteal artery, in the target limb confirmed at baseline. (Note: treatment of outflow disease is permitted. Drug-eluting devices are not allowed for outflow treatment)

Exclusion Criteria:

1. Females who are pregnant, lactating, or intended to become pregnant, or males intending to father children during the study
2. Subject under current medication known to affect CYP3A4 metabolism, or consuming food or beverages that are known substrates of CYP3A4
3. Contraindication to dual anti-platelet therapy
4. Subject receiving chronic anticoagulation therapy (e.g. low molecular weight heparin, warfarin, or novel direct oral anticoagulants (N(D)OACs)) if the treatment cannot be interrupted 48 hours prior to the procedure
5. Known intolerance to study medications, Limus- like drug or contrast agents that in the opinion of the investigator could not be adequately pretreated
6. Current participation in an investigational drug or another device study
7. History of hemorrhagic stroke within 3 months
8. Patients with a history of Myocardial Infarction (MI) or thrombolysis within 30 days prior-index procedure
9. Previous or planned surgical or interventional procedure within 14 days before or 30 days after index procedure (successful treatment of the ipsilateral and contralateral iliac arteries is permitted during the index procedure. Drug-eluting devices are not allowed for treatment of the occluded inflow iliac arteries)
10. Prior endovascular treatment of the target lesion (e.g., POBA, DCB, BMS, DES, cutting balloons, scoring balloons, cryoplasty, thrombectomy, atherectomy, brachytherapy or laser devices)
11. Previous placement of a bypass graft proximal to the target lesion
12. Chronic renal insufficiency (eGFR < 30 mL/min within 72 hours prior to index procedure)
13. Patient requiring renal replacement therapy
14. No normal proximal arterial segment in which duplex ultrasound velocity ratios could be measured.
15. Subject is unable to walk without assistance (e.g. walker, cane).
16. Subject is receiving immunosuppressant therapy.
17. Subject has known or suspected active infection at the time of the index procedure.
18. Subject has platelet count < 100,000/mm3 or > 700,000/mm3.
19. Subject has white blood cell (WBC) count < 3,000/mm3.
20. Subject is unable to tolerate blood transfusions because of religious beliefs or other reasons.
21. Subject has history of gastrointestinal hemorrhage requiring a transfusion within 3 months prior to the index procedure.
22. Life expectancy less than 12 months due to other comorbidities, that in the investigators opinion, could limit subject ability to comply with the study required follow-up visits/procedure and threaten the study scientific integrity
23. Treatment of the contralateral limb during the same procedure or within 30 days following the study procedure (exclusive of the iliac arteries, which can be treated during the index procedure if no drug eluting technology is used)
24. Non femoral vascular access
25. Target lesion would require treatment with more than two BRight balloons
26. Known inadequate distal outflow
27. Acute or sub-acute thrombus in the target vessel
28. Aneurysmal target vessel
29. Use of adjunctive therapies (i.e. laser, atherectomy, cryoplasty, scoring/cutting balloon, brachytherapy) during the study procedure in the target lesion or target vessel
30. Presence of concentric calcification that precludes PTA pre-dilatation
31. Significant contralateral or ipsilateral common femoral disease that requires intervention during the index procedure
32. Persistent hemodynamically-significant stenosis following predilatation or residual stenosis of >30%, stent placement, or flow-limiting (Grade D or greater) dissection following pre-dilatation
33. In-stent restenosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-06-27 (Actual); Study Completion 2025-07-22 (Actual)

PRIMARY OUTCOMES:
AUC 0-t | 0 to 24 hours
  Area under the drug concentration-time curve, calculated using linear trapezoidal summation from time zero to time tlast, where tlast is the time of the last measurable concentration (Ct).
AUC 0-inf | 0 to 24 hours
  Area under the drug concentration-time curve from time zero to infinity
Cmax | 0 to 24 hours
  Maximum observed drug concentration
Terminal Elimination Rate Constant (λz) | 0 to 24 hours
  Apparent terminal elimination rate constant, calculated by linear regression of the terminal linear portion of the log concentration vs. time curve
Terminal Elimination Half-life (t1/2) | 0 to 24 hours
  Apparent terminal elimination half-life, calculated as ln(2)/λz
tmax | 0 to 24 hours
  Time of the maximum drug concentration (obtained without interpolation). If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value.
Drug clearance (CL) | 0 to 24 hours
  Apparent total clearance, calculated as dose/AUC0-inf
Apparent volume of distribution at the terminal phase (Vz) | 0 to 24 hours
  Apparent volume of distribution at the terminal phase, calculated as CL/λz
Metabolic Ratio (MR) | 0 to 24 hours
  Metabolic ratio calculated as the molar concentration of sirolimus AUC0-inf to BIOtorcin AUC0-inf

SECONDARY OUTCOMES:
Device success | during procedure
  Successful delivery, balloon inflation/deflation and retrieval of the intact trial device
Acute technical success | during procedure
  Successful vascular access and completion of the endovascular procedure and immediate achievement of a final residual diameter stenosis of ≤30% of the treated lesion by core laboratory assessed QVA on the completion angiography with no bailout stenting
Acute procedural success | 72 hours post procedure
  Technical success without the occurrence of death, major target limb amputation, thrombosis of the target lesion, or clinically-driven TLR within 72 hours of the index procedure
Major adverse event (MAE) rate | 1, 6 and 12 months post index procedure
  MAE is a composite of device or procedure related death within 30 days post index procedure, or major index limb amputation, or cd TLR at 1, 6 and 12 months post index procedure
Clinically-driven Target Lesion Revascularization (cd TLR) rate | 1, 6 and 12 months post index procedure
  cd TLR is defined as any repeat intervention of the target lesions or surgical bypass of the target vessel performed for restenosis > 50% or other complication involving the target lesion, after documentation of recurrent clinical symptoms of the patient.
Clinically-driven Target Vessel Revascularization (cd TVR) rate | 1, 6 and 12 months post index procedure
  cd TVR, defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel, after documentation of recurrent clinical symptoms of the patient.
All-cause of death rate | 1, 6 and 12 months post index procedure
Target limb major (above the ankle) and minor (below the ankle) amputation rate | 1, 6 and 12 months post index procedure
Change in Rutherford Classification as compared to baseline | 1, 6 and 12 months post index procedure
Change in Ankle Brachial Index (ABI) as compared to baseline | 1, 6 and 12 months post index procedure
Change in Walking Impairment Questionnaire (WIQ) as compared to baseline | 1, 6 and 12 months post index procedure
Target lesion Binary Restenosis rate | 1, 6 and 12 months post index procedure
  Defined as duplex ultrasound peak systolic velocity ratio (PSVR) > 2.5 or angiographic assessment which suggests stenosis > 50% by QVA
Target lesion Primary Patency rate | 1, 6 and 12 months post index procedure
  Defined as duplex ultrasound peak systolic velocity ratio (PSVR) ≤ 2.5 or angiographic assessment which suggests stenosis ≤ 50% by QVA and the absence of Clinically-driven TLR (adjudicated by a CEC)
embolic event of the index limb rate | during procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Perth Hospital, Perth, WAUS, Australia

IPD SHARING:
Plan to Share IPD: No